CLINICAL TRIAL: NCT04967469
Title: Comparison of Serum Calcium Level Between Preoperative Vitamin D and Non-vitamin D Regimen of Total Parathyroidectomy in End-stage Renal Failure Patients in Rajavithi Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 63127
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2021-08

CONDITIONS: End Stage Renal Disease
Keywords: Hypocalcemia; Hyperparathyroidism; End Stage Renal Disease (ESRD); calcitriol
MeSH Terms: conditions — Kidney Failure, Chronic; Hypocalcemia; Hyperparathyroidism | interventions — Calcitriol; alfacalcidol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- take calcitriol (Experimental): End-stage renal failure patients who is Hyperparathyroid with ESRD take calcitriol
  Interventions: Drug: Calcitriol
- take alphacalcidol (Experimental): End-stage renal failure patients who is Hyperparathyroid with ESRD take 1-hydroxycholecalciferol (alfacalcidol)
  Interventions: Drug: Alfacalcidol 0.5 MCG Oral Capsule
- control (No Intervention): End-stage renal failure patients who is Hyperparathyroid with ESRD take standard treatment

INTERVENTIONS:
Drug: Calcitriol — end-stage renal failure patients who is hyperparathyroid with ESRD take calcidol preoperative Parathyroidectomy
  Arms: take calcitriol
Drug: Alfacalcidol 0.5 MCG Oral Capsule — end-stage renal failure patients who is hyperparathyroid with ESRD take alfacalcidol preoperative Parathyroidectomy
  Arms: take alphacalcidol

SUMMARY:
This Research is compare about IV Calcium between end-stage renal failure patients who take vitamin D and non-vitamin D preoperative parathyroidectomy

ELIGIBILITY:
Inclusion Criteria:

* New End-stage renal failure patients and have iPTH>800 pg/dl at least 6 months
* Patients who no response hyperphosphatemia with high dose vitamin D

Exclusion Criteria:

* Allergy vitamin D
* Pregnancy
* Patients who parathyroidectomy have less than 4 gland

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of serum calcium level between patients who take Vitamin D and non-Vitamin D | 4 year
  Comparison of serum calcium level between patients who take Vitamin D and non-Vitamin D

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No